CLINICAL TRIAL: NCT06334848
Title: Efficacy of Mini Sling Versus Transobturator Tape in Surgical Management of Women With Stress Urinary Incontinence
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Tarek Salem Rezk, Principal Investigator, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TOT versus mini sling
Record Dates: First submitted 2024-03-12; First posted 2024-03-28 (Actual); Last update posted 2024-03-28 (Actual); Status verified 2024-03

CONDITIONS: Stress Urinary Incontinence
MeSH Terms: conditions — Urinary Incontinence, Stress | interventions — Suburethral Slings

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- treatment of stress urinary incontinence by transobturator tape (Other): patients with stress urinary incontinence are treated by transobturator tape
  Interventions: Procedure: transobturator tape
- treatment of stress urinary incontinence by mini sling (Other): patients with stress urinary incontinence are treated by mini sling
  Interventions: Procedure: transobturator tape

INTERVENTIONS:
Procedure: transobturator tape — Women with stress urinary incontinence are treated by transobturator tape versus mini sling
  Other Names: mini sling

SUMMARY:
To compare the efficacy of mini sling against Transobturator tape for surgical management of women with stress urinary incontinence.

DETAILED DESCRIPTION:
Urinary incontinence is defined as involuntary loss of urine and is divided into subtypes according to symptoms. These subtypes include SUI, in which urine loss occurs during exertion, physical exercise, coughing or sneezing; urgency urinary incontinence (UUI), in which urine loss is associated with urinary urgency; and mixed urinary incontinence (MUI), which is characterized by the association of stress loss with urgency.

There are non-surgical treatments (e.g., lifestyle modifications, pharmacotherapy, physiotherapy and vaginal pessary) and surgical treatments.

As regards sling use, it was found that mid urethral slings techniques achieved high cure rates in women with SUI and have become the mainstay for surgical treatment of SUI in women over the last 2 decades.

One of the modalities of such procedures is the transobturator mid urethral tape (TOT). It was introduced to minimize the complications of the previous retropubic tapes, which include injury to the bladder, major vessels, and bowel.

In an effort to maintain efficacy while eliminating some of the side effects, a new generation of tapes has been developed, called single incision tapes or mini-slings. They are designed to be shorter in length than standard mid-urethral slings and do not penetrate the tissues as deeply as standard slings.

ELIGIBILITY:
Inclusion Criteria:

* Women with a medical history of SUI
* mixed urinary incontinence (MUI) in which SUI had to be the dominating symptom
* confirmed by a positive standardized cough test with 300 cm3 water in the bladder

Exclusion Criteria:

* Women will be excluded if they are aged >60 years
* had previous incontinence or pelvic organ prolapse surgery
* planned or present pregnancy
* residual urine volume>100 ml
* previous pelvic irradiation
* neurological conditions such as multiple sclerosis
* current treatment with corticoids
* history of genital or abdominal cancer or a pelvic mass.

Max Age: 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 42 (Estimated)
Dates: Start 2024-04 (Estimated); Primary Completion 2025-04 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Comparing Mini Sling and Transobturator Tape in Surgical Management of Women with Stress Urinary Incontinence regarding incidence of complications | one year
  comparing between mini sling and transobturator tape in surgical management of women with stress urinary incontinence regarding:
  • Urinary continence measured by ICIQ(international continence index questionnaire)
Comparing Mini Sling and Transobturator Tape in Surgical Management of Women with Stress Urinary Incontinence regarding postoperative pain | one year
  comparing between mini sling and transobturator tape in surgical management of women with stress urinary incontinence regarding:
  • Post operative pain measured by NRS(numerical rating pain score)

SECONDARY OUTCOMES:
Comparing Mini Sling and Transobturator Tape in Surgical Management of Women with Stress Urinary Incontinence regarding sexual function | one year
  comparing between mini sling and transobturator tape in surgical management of women with stress urinary incontinence regarding:
  • Sexual function measured by FSFI(female sexual function index)

REFERENCES:
- [Background] D'Ancona C, Haylen B, Oelke M, Abranches-Monteiro L, Arnold E, Goldman H, Hamid R, Homma Y, Marcelissen T, Rademakers K, Schizas A, Singla A, Soto I, Tse V, de Wachter S, Herschorn S; Standardisation Steering Committee ICS and the ICS Working Group on Terminology for Male Lower Urinary Tract & Pelvic Floor Symptoms and Dysfunction. The International Continence Society (ICS) report on the terminology for adult male lower urinary tract and pelvic floor symptoms and dysfunction. Neurourol Urodyn. 2019 Feb;38(2):433-477. doi: 10.1002/nau.23897. Epub 2019 Jan 25. PMID 30681183
- [Background] Khandelwal C, Kistler C. Diagnosis of urinary incontinence. Am Fam Physician. 2013 Apr 15;87(8):543-50. PMID 23668444
- [Background] Leslie SW, Tran LN, Puckett Y. Urinary Incontinence. 2024 Aug 11. In: StatPearls [Internet]. Treasure Island (FL): StatPearls Publishing; 2025 Jan-. Available from http://www.ncbi.nlm.nih.gov/books/NBK559095/ PMID 32644521
- [Background] Falah-Hassani K, Reeves J, Shiri R, Hickling D, McLean L. The pathophysiology of stress urinary incontinence: a systematic review and meta-analysis. Int Urogynecol J. 2021 Mar;32(3):501-552. doi: 10.1007/s00192-020-04622-9. Epub 2021 Jan 8. PMID 33416968
- [Background] Kowalik CG, Dmochowski RR, De EJB. Surgery for female SUI: The ICI algorithm. Neurourol Urodyn. 2019 Aug;38 Suppl 4:S21-S27. doi: 10.1002/nau.23879. Epub 2019 May 2. PMID 31050030
- [Background] Novara G, Ficarra V, Boscolo-Berto R, Secco S, Cavalleri S, Artibani W. Tension-free midurethral slings in the treatment of female stress urinary incontinence: a systematic review and meta-analysis of randomized controlled trials of effectiveness. Eur Urol. 2007 Sep;52(3):663-78. doi: 10.1016/j.eururo.2007.06.018. Epub 2007 Jun 21. PMID 17601652
- [Background] Kim A, Kim S, Kim HG. Current Overview of Surgical Options for Female Stress Urinary Incontinence. Int Neurourol J. 2020 Sep;24(3):222-230. doi: 10.5213/inj.2040052.026. Epub 2020 Sep 30. PMID 33017893
- [Background] Nambiar A, Cody JD, Jeffery ST, Aluko P. Single-incision sling operations for urinary incontinence in women. Cochrane Database Syst Rev. 2017 Jul 26;7(7):CD008709. doi: 10.1002/14651858.CD008709.pub3. PMID 28746980
- [Background] Cox A, Herschorn S, Lee L. Surgical management of female SUI: is there a gold standard? Nat Rev Urol. 2013 Feb;10(2):78-89. doi: 10.1038/nrurol.2012.243. Epub 2013 Jan 15. PMID 23318365
- [Background] Rudnicki M, von Bothmer-Ostling K, Holstad A, Magnusson C, Majida M, Merkel C, Prien J, Jakobsson U, Teleman P. Adjustable mini-sling compared with conventional mid-urethral slings in women with urinary incontinence. A randomized controlled trial. Acta Obstet Gynecol Scand. 2017 Nov;96(11):1347-1356. doi: 10.1111/aogs.13205. Epub 2017 Sep 15. PMID 28815547
- [Background] Emami M, Momtazan A, Maghsoudi R, Ameli M, Kashi A, Amirpoor M, Karimi S. Transobturator tape and mini-sling methods in stress urinary incontinence: Results of a randomized clinical trial. Urologia. 2019 Aug;86(3):152-155. doi: 10.1177/0391560319845255. Epub 2019 May 10. PMID 31072274
- [Background] Chang CP, Chang WH, Hsu YM, Chen YJ, Wen KC, Chao KC, Yen MS, Horng HC, Wang PH; Task Force on Gyn-Urodynamic Research Group. Comparison of single-incision mini-slings (Ajust) and standard transobturator midurethral slings (Align) in the management of female stress urinary incontinence: A 1-year follow-up. Taiwan J Obstet Gynecol. 2015 Dec;54(6):726-30. doi: 10.1016/j.tjog.2015.10.007. PMID 26700993
- [Background] Kokanali MK, Doganay M, Aksakal O, Cavkaytar S, Topcu HO, Ozer I. Risk factors for mesh erosion after vaginal sling procedures for urinary incontinence. Eur J Obstet Gynecol Reprod Biol. 2014 Jun;177:146-50. doi: 10.1016/j.ejogrb.2014.03.039. Epub 2014 Apr 13. PMID 24793930
- [Background] Maturana AP, Palos CC, Ghersel FR, Fernandes CE, Oliveira E. Randomized controlled trial comparing mini-sling with transobturator sling for the treatment of stress urinary incontinence. Int Urogynecol J. 2020 Sep;31(9):1925-1931. doi: 10.1007/s00192-019-04145-y. Epub 2019 Nov 29. PMID 31784809